CLINICAL TRIAL: NCT04023825
Title: Analgesic Contribution of the Suprazygomatic Maxillary Nerve Block for Cleft Palate Surgery in Children
Acronym: Suprazyg
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no participants enrolled
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI2018_843_0020
Record Dates: First submitted 2019-07-16; First posted 2019-07-18 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Cleft Palate; Surgery
Keywords: cleft palate; surgery; maxillary nerve block; local anesthetic; loco regional anesthesia; face nerve block
MeSH Terms: conditions — Cleft Palate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Patients will receive loco regional anesthesia
  Interventions: Drug: suprazygomatic maxillary nerve block
- control group (No Intervention): Patients will not receive loco regional anesthesia

INTERVENTIONS:
Drug: suprazygomatic maxillary nerve block — in the experimental group, each child will profit from the realization of a suprazygomatic maxillary nerve block.
  Arms: experimental group

SUMMARY:
This is a monocentric prospective randomized simple-blind designed study evaluating the superiority of the suprazygomatic maxillary nerve block in analgesia after cleft palate surgery compared with a control group. Every two hours, nurses systematically reassess the patient's pain and adjust the analgesic medications. Analgesic requirement, incidence of respiratory complications, re-feeding time and the duration of hospitalization are evaluated.

DETAILED DESCRIPTION:
Cleft palate is the most common congenital malformation and requires early surgery given the complications it generates. The surgical site involving the upper airways and the use of morphine are providers of respiratory complications. The suprazygomatic maxillary nerve block could considerably reduce the use of morphine in the postoperative period and thus the respiratory complications in addition to an optimal comfort for the patient. The primary endpoint was to evaluate morphine consumption during the first postoperative 48 hours after cleft palate surgery.

ELIGIBILITY:
Inclusion Criteria:

* children between 5 months and 12 years old
* weight >5kg
* children undergoing cleft palate repair surgery with or without upper lip surgery

Exclusion Criteria:

* inappropriate age
* weight <5kg
* abnormal blood coagulation
* local anesthetic contraindication (including levobupivacaine, as well as any other associated treatment administered in this clinical study, including opioids, general anesthetics such as ketamine or propofol, paracetamol or corticosteroids)
* local infection

Ages: 5 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline of morphine consumption | up to 48 hours after cleft palate surgery
  The main objective of this study is to compare the consumption of morphine during the first 48 hours after cleft palate surgery in a group of patients treated by realization of a suprazygomatic maxillary nerve block, compared to a control group.

SECONDARY OUTCOMES:
Change from baseline of consumption of perioperative morphine | up to one week after cleft palate surgery
  evaluation of the consumption of perioperative morphine
Measure of the number of episodes of respiratory distress | up to one week after cleft palate surgery
  Measure of the number of episodes of respiratory distress
Measure of the period of re-feeding | up to one week after cleft palate surgery
  Measure of the period of re-feeding
Measure of the duration of hospitalization | up to one week after cleft palate surgery
  Measure of the duration of hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Matthieu Miclo, MD, Principal Investigator — CHU Amiens; Emmanuel Lorne, Pr, Principal Investigator — CHU Amiens; Jérémie Garnier, MD, Principal Investigator — CHU Amiens; Marie Trujillo-Garcia, MD, Principal Investigator — CHU Amiens; Dimitri Santarelli, MD, Principal Investigator — CHU Amiens; Cica Carole Gbaguidi, MD, Principal Investigator — CHU Amiens

IPD SHARING:
Plan to Share IPD: No